CLINICAL TRIAL: NCT02625402
Title: Pilot RCT Comparing Effectiveness of Two Decision Aids for Hip and Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Newton-Wellesley Hospital (Other)
Responsible Party: Principal Investigator, Karen Sepucha, Associate Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2013P001794
Record Dates: First submitted 2015-12-04; First posted 2015-12-09 (Estimated); Results first posted 2017-12-18 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-09

CONDITIONS: Hip Osteoarthritis; Knee Osteoarthritis
Keywords: decision making; decision aids; decision quality instruments; osteoarthritis; shared decision making
MeSH Terms: conditions — Osteoarthritis, Hip; Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interactive decision aid (Experimental): Group receiving brief interactive decision aid. The decision aids are the Shared Decision Points for hip and knee osteoarthritis from Healthwise
  Interventions: Behavioral: Brief interactive decision aid
- Video decision aid (Experimental): Group receiving long video decision aids. The decision aids are the hip or knee DVD and Booklets for hip and knee osteoarthritis from Health Dialog
  Interventions: Behavioral: Long video decision aid

INTERVENTIONS:
Behavioral: Brief interactive decision aid — The Healthwise Shared Decision Points in booklet version for hip and knee osteoarthritis
  Arms: Interactive decision aid
Behavioral: Long video decision aid — Health Dialog DVD and booklet decision aids for hip and knee osteoarthritis
  Arms: Video decision aid

SUMMARY:
This pilot RCT study is to examine the comparative effectiveness of two decision aids for hip and knee osteoarthritis.

DETAILED DESCRIPTION:
This pilot RCT study is to examine the comparative effectiveness of two decision aids for hip and knee osteoarthritis. The vendors employ different design features (e.g. use of video for patient narratives, interactive values clarification exercise) and the study will examine the relative impact of the different features on decision quality. Eligible subjects will be randomly assigned to receive one of two decision aids before their upcoming clinic visit with a participating provider. Immediately before the visit, participants will complete a short questionnaire about the decision aid. This pilot study will assist with determining the potential difference between these two decision aids on improving knowledge and use of decision aids.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of either hip or knee osteoarthritis
* Scheduled visit with participating orthopedic surgeon

Exclusion Criteria:

* Prior partial or total knee or hip replacement surgery
* Hip fracture or aseptic necrosis in the last 12 months
* Rheumatoid arthritis or psoriatic arthritis
* Unable to read or speak English

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen R Sepucha, PhD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Newton Wellesley Hospital, Newton, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sepucha K, Feibelmann S, Chang Y, Clay CF, Kearing SA, Tomek I, Yang T, Katz JN. Factors associated with the quality of patients' surgical decisions for treatment of hip and knee osteoarthritis. J Am Coll Surg. 2013 Oct;217(4):694-701. doi: 10.1016/j.jamcollsurg.2013.06.002. Epub 2013 Jul 25. PMID 23891070
- Available data/document: Outcome measure — https://mghdecisionsciences.org/tools-training/decision-quality-instruments/ — Hip Osteoarthritis Decision Quality Instrument
- Available data/document: Outcome measure — https://mghdecisionsciences.org/tools-training/decision-quality-instruments/ — Knee Osteoarthritis Decision Quality Instrument

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient recruitment was conducted from December 2015 to March 2016. Patients were recruited at two hospitals. Consent for the study (or enrollment) was implied by completion of the survey, so the enrollment number is lower than the number that started the study and were assigned to a study arm.
Period: Overall Study
Arm/Group | Interactive Decision Aid | Video Decision Aid
Started | 42 | 37
Completed | 33 | 25
Not Completed | 9 | 12

BASELINE CHARACTERISTICS:
Population: The study participants between both groups were quite balanced. Mean age and gender did not have any significant differences based on group assignment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Interactive Decision Aid | Video Decision Aid | Total
Number analyzed (Participants) | 33 | 25 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.3 (8.7) | 62.8 (8.5) | 63.7 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants] — Gender data was collected through chart review of enrolled patients.
  Participants
    Female | 16 | 14 | 30
    Male | 17 | 11 | 28
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Hip and Knee Decision Quality Instruments Knowledge Subscale Scores
Description: 5 multiple choice knowledge items from the Hip and Knee Decision Quality Instruments will be averaged into a knowledge subscale score (0-100%) with higher scores indicating higher knowledge.
Time Frame: In clinic, immediately before the first visit with surgeon
Population: The total knowledge score of 5 multiple questions with a total score of 0-100% was generated for all study patients.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Interactive Decision Aid | Video Decision Aid
Number analyzed (Participants) | 33 | 25
units on a scale | 55.2 (25.5) | 48.8 (32.2)
Statistical Analysis 1: Comparison: Interactive Decision Aid vs Video Decision Aid; Test type: Equivalence — Knowledge scores within 10% points; p < 0.05, t-test, 2 sided; Mean Difference (Final Values) = 6.4, 95% CI 2-sided [-8.8 to 21.5], Standard Error of Mean 7.6

2. Secondary Outcome: Percentage of Participants Who Used the Decision Aid
Description: 1 item asking patients how much they reviewed the program (none, some. most, all). The percentage who report viewing most or all will be calculated.
Time Frame: In clinic, immediately before the first visit with surgeon
Population: We wanted to assess how much patients reviewed whichever decision aid they were randomized to before their visit. As such, we assessed how much they reviewed of the program (none, some, most, all) and will share the categorical results.
Measure: Count of Participants; unit: Participants
Arm/Group | Interactive Decision Aid | Video Decision Aid
Number analyzed (Participants) | 33 | 25
Participants
  Reviewed most or all of the DA | 23 | 14
  Reviewed none or some of the DA | 8 | 11
  Missing | 2 | 0

3. Secondary Outcome: Percentage of Participants With a Clear Treatment Preference
Description: 1 item assessing patient's treatment preference (surgery, non-surgical options, or not sure). The percentage who have a clear preference (either for surgery or non surgical options) will be calculated.
Time Frame: In clinic, immediately before the first visit with surgeon
Measure: Count of Participants; unit: Participants
Arm/Group | Interactive Decision Aid | Video Decision Aid
Number analyzed (Participants) | 33 | 25
Participants
  Clear preference | 22 | 15
  Not sure | 11 | 10

ADVERSE EVENTS:
Time Frame: Serious and other (not including serious) adverse events were not collected/assessed.
Description: Adverse events were not collected as part of this survey study.
Arm/Group | Interactive Decision Aid | Video Decision Aid
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No